CLINICAL TRIAL: NCT00979069
Title: Aerobic Exercise to Improve Executive Language Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E6860-M
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Group (Experimental): 12 weeks of aerobic exercise 3 times a week
  Interventions: Behavioral: Aerobic group
- Control Group (No Intervention): No contact control

INTERVENTIONS:
Behavioral: Aerobic group — 12 weeks of aerobic exercise 3 times a week
  Arms: Aerobic Group

SUMMARY:
The purpose of this study is to see if exercise can improve brain function in older adults

DETAILED DESCRIPTION:
Recently, considerable attention has been devoted to examining the beneficial relationship between cognition and aerobic exercise in older adults. Specifically, the effects are thought to involve higher order cognitive processes, such as working memory, switching between tasks, and inhibiting irrelevant information, all of which are thought to be sub- served, in part, by the frontal lobes (Colcombe et al., 2006). Importantly, these areas also are most susceptible to age-related decline (Raz, 2000) and are essential resources for language production (Kemper & Sumner, 2001; Murray & Lenz, 2001). However, despite promising cognitive improvement, changes in frontally-mediated executive language functions have been widely ignored. This is unfortunate considering impaired word retrieval compromises communicative effectiveness, leading to frustration, depression, and withdrawal. Perhaps more importantly, communication ineffectiveness, particularly in the elderly, leads to difficulties interacting with health care professionals leading to further health care burdens. Since cognition, and specifically word retrieval difficulties, usually remain untreated, it is important to find treatment strategies for minimizing these deficits. Therefore, the short-term goal and the purpose of this proposal is to examine the potential of aerobic exercise to improve executive language function in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Consent of participants' primary health care physicians to participate in the aerobic exercise.
* Patients must not have participated in any consistent exercise program or experimental study for at least 3 months prior to enrollment.
* They must be capable of providing informed consent and complying with the trial procedures.

Exclusion Criteria:

* Demented as defined by the Modified Mini Mental Status Exam.
* Unalterable travel schedules.
* Site accessibility constraints.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe R Nocera, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (2):
- United States (2):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia

REFERENCES:
- [Result] Nocera JR, McGregor KM, Hass CJ, Crosson B. Spin exercise improves semantic fluency in previously sedentary older adults. J Aging Phys Act. 2015 Jan;23(1):90-4. doi: 10.1123/japa.2013-0107. Epub 2014 Jan 14. PMID 24425525

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Group | Control Group
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Group | Control Group | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 8 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 6 | 4 | 10
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Executive Language Functions
Description: The Verbal Fluency Test is demonstrated to be reliable and valid among adults aged 50 to 89 (Delis, et al., 2001; Delis, Kramer, Kaplan, & Hodnack, 2004). The Verbal Fluency Test has three conditions, Letter Verbal Fluency, Category Verbal Fluency, and Switching Verbal Fluency. Each was randomized at pre- and post-12 week timeline and equated for difficulty. Letter Verbal Fluency assesses the number of words beginning with certain letters that participants can generate within 60 seconds,the Category Verbal Fluency assesses the number of words within particular categories participants can generate within 60 seconds, and the Switching Verbal Fluency assesses the number of words while alternating between different categories participants can generate within 60 seconds. For each condition (letter, category, and switching) a total score representing the total number of correct
Time Frame: number of correct words at pre and post separated by 12 weeks
Measure: Mean (Standard Deviation); unit: Mean outpoint by group at pre and post
Arm/Group | Aerobic Group | Control Group
Number analyzed (Participants) | 10 | 8
Mean outpoint by group at pre and post
  Letter Verbal Fluency- Pre | 31.6 (6.0) | 30.8 (3.6)
  Letter Verbal Fluency- Post | 33.7 (6.0) | 31.8 (2.6)
  Category Verbal Fluency- Pre | 39 (5.4) | 40.2 (3.9)
  Category Verbal Fluency- Post | 45.1 (8.1) | 41 (4.4)
  Switching Verbal Fluency- Pre | 10.6 (2.5) | 11.4 (1.7)
  Switching Verbal Fluency- Post | 13.1 (1.7) | 12.8 (2.5)

ADVERSE EVENTS:
Time Frame: During study collection
Arm/Group | Aerobic Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No